CLINICAL TRIAL: NCT00601159
Title: Phase Ⅱ Study of Gemcitabine and Cisplatin as First Line Combination Therapy in Patients With Triple-negative MBC
Brief Title: Gemcitabine and Cisplatin as First Line Combination Therapy in Patients With Triple-negative MBC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Base for drug clinical trials, Fudan University cancer hospital, Fudan University cancer hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200709GP
Record Dates: First submitted 2007-12-26; First posted 2008-01-25 (Estimated); Last update posted 2011-07-04 (Estimated); Status verified 2011-06

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer; triple-negative Breast Cancer; cisplatin; chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gemcitabine and cisplatin (Experimental): cisplatin and gemcitabine in the management of triple negative metastatic breast cancer
  Interventions: Drug: gemcitabine and cisplatin

INTERVENTIONS:
Drug: gemcitabine and cisplatin — Cispaltin 25mg/m2，ivgtt，D1, 2, 3 gemcitabine 1000mg/m2，ivgtt，30'，D1, 8 repeat every 3 weeks
  Other Names: gemzar

SUMMARY:
Primary objective of this study is to evaluate the efficacy of gemcitabine and cisplatin as first line therapy in patients with triple-negative MBC. 80 patients will be treated into this study.

DETAILED DESCRIPTION:
Triple-negative breast tumors could contribute to the poor prognosis comparing with luminal A breast cancer.Fewer study has revealed that Cisplatin-based therapy may be effective for this type breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Give written informed consent prior to study, with understanding that the patient has the right to withdraw from the study at any time without prejudice
* Be female and ≥18 and ≤75 years of age
* Be ambulatory and have ECOG performance stastus of ≤1
* Have histological confirmed breast cancer,and the speciman confirmed ER negative,PR negatiev, and HER-2 negative by immunochemistry technich of Fudan cancer hospital.
* Locally advanced or metastastic breast cancer who didn't receive first-line chemotherapy. No matter whether the patient has received anthracyclin or taxane treatment as neo-adjuvant or adjuvant treatment.
* Have at least one target lesion according to the RECIST criteria.

Exclusion criteria:

* Preganant or lactating women
* Advaced patient has received one or more chemotherapies
* Chemotherapy within four weeks preceding treatment start
* ECOG ≥ 2
* Radiotherapy to the axial skeleton within the 4 weeks preceding study treatment start or insufficient recovery from the effects of prior radiotherapy
* Participation in any investigational drug study within 4 weeks preceeding treatment start
* Evidence of CNS metastasis
* History of another malignacy within the last five years except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix or a contralateral breast cancer
* Abnormal laboratory values: hemoglobin < 8. 0g/dl, neutrophil< 1.5×109/L, platelet< 100×109/L.
* serum creatine > upper limit of normal (ULN)
* serum bilirubin > ULN
* ALT and AST >5×ULN
* AKP >5×ULN
* Serious uncontrolled intercurrence infection
* Life expectancy of less than 3 months

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-09; Primary Completion 2010-05 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
PFS (progression free survival) | 1 year

SECONDARY OUTCOMES:
side effects | 6 months
BRCA1 mutation realtionship with efficacy and toxicity analysis | at the end of therapy
pharmacogenetic analysis | collect blood samples before therapy

CONTACTS AND LOCATIONS:
Overall Officials: Zhonghua Wang, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Turner NC, Reis-Filho JS, Russell AM, Springall RJ, Ryder K, Steele D, Savage K, Gillett CE, Schmitt FC, Ashworth A, Tutt AN. BRCA1 dysfunction in sporadic basal-like breast cancer. Oncogene. 2007 Mar 29;26(14):2126-32. doi: 10.1038/sj.onc.1210014. Epub 2006 Oct 2. PMID 17016441
- [Derived] Zhang J, Wang Z, Hu X, Wang B, Wang L, Yang W, Liu Y, Liu G, Di G, Hu Z, Wu J, Shao Z. Cisplatin and gemcitabine as the first line therapy in metastatic triple negative breast cancer. Int J Cancer. 2015 Jan 1;136(1):204-11. doi: 10.1002/ijc.28966. Epub 2014 May 23. PMID 24824628